CLINICAL TRIAL: NCT04244851
Title: Nutritional State and Care Pathway of Hospitalized Malnourished Patients, Within 3 Months of Admission
Acronym: Nutriker
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC19_30034_NUTRIKer; 2019-A01809-48 (Other: ansm)
Record Dates: First submitted 2019-12-13; First posted 2020-01-28 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-01

CONDITIONS: Malnutrition
Keywords: Malnutrition,; qualitative study
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Malnourished patients: Malnourished patients
  Interventions: Other: Malnourished patients

INTERVENTIONS:
Other: Malnourished patients — Data of included patients will be recorded during hospitalization using medical charts.
  Every patient will be contacted by phone 3 months after hospital discharge. A sample of patients and their caregivers will be interviewed to better understand their perception of malnutrition and what they need to better take care of malnutrition.

SUMMARY:
Malnourished patients are at risk of many complications, including infections, pressure ulcers and readmissions. Little is known about their care pathway after hospital discharge.

This study aims to determine care pathways of malnourished patients after hospital discharge and to determine what they need to better take care of their malnutrition.

DETAILED DESCRIPTION:
All patients hospitalized in the post-emergency unit of Rennes University Hospital during the study period will be screened for malnutrition.

Data concerning newly diagnosed malnourished patients will be recorded and those patients will be contacted 3 months after their hospital discharge.

A qualitative study will be conducted among malnourished patients and their families : a sample of patients and their caregivers will be interviewed to better understand their perception of malnutrition and what they need to better take care of malnutrition.

ELIGIBILITY:
Inclusion Criteria:

* Malnourished patients, hospitalized in the post-emergency unit during the study period, according to the malnutrition diagnostic criteria defined by the French Health Authority :
* age ≥ 70 years old: weight loss ≥ 5% within 1 month or ≥ 10% within 6 months and/or BMI <21 and or serum albumin level < 35 g/l
* age < 70 years old : weight loss ≥ 5% in 1 month or ≥ 10% in 6 months or ≥ 10% compared to the usual weight before the onset of the disease; or BMI <18.5 kg / m2

Non-inclusion criteria :

* refusing to participate in the study
* age < 18 years old
* patients under tutorship or guardianship
* patients living in retirement home
* Patients without a fixed address

Exclusion criteria :

-patients transferred in another unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Malnourished patients diagnosed during their hospitalization in the post-emergency unit of Rennes Universisty Hospital
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-02-04 (Actual); Primary Completion 2020-10-04 (Estimated); Study Completion 2020-10-04 (Estimated)

PRIMARY OUTCOMES:
evolution of malnutrition after hospital discharge | 3 months after discharge
  Malnutrition diagnostic criteria defined by the French Health Authority :
  * If age ≥ 70 years old : weight loss ≥ 5% within 1 month and/or ≥ 10% within 6 months and/or BMI < 21 kg/m² and/or serum albumin level < 35 g/l
  * If age < 70 years old: weight loss ≥ 5% within 1 month and/or ≥ 10% within 6 months and/or BMI < 18,5 kg/m² level

SECONDARY OUTCOMES:
Describe the path of care following the hospitalization of patients diagnosed with malnutrition at the hospital | 3 months after discharge
  * Number of hospital readmissions
  * Number of family physician consultations
Evaluate appropriation of patient regarding malnutrition | 3 months after discharge
  Qualitative study by semi-structured patient interviews
Evaluate the perception of patient regarding malnutrition | 3 months after discharge
  Qualitative study by semi-structured patient interviews
Evaluate expectations of patient regarding malnutrition | 3 months after discharge
  Qualitative study by semi-structured patient interviews
Evaluate the needs of health professionals regarding undernutrition | 3 months after discharge
  Qualitative study by semi-structured patient interviews
Evaluate the expectations of health professionals regarding undernutrition | 3 months after discharge
  Qualitative study by semi-structured patient interviews
Evaluate knowledge of health professionals regarding undernutrition | 3 months after discharge
  Qualitative study by semi-structured patient interviews

CONTACTS AND LOCATIONS:
Locations (1):
- Rennes University Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided